CLINICAL TRIAL: NCT07302724
Title: Drain Removal Before Versus After Continuous Passive Motion in Primary Total Knee Arthroplasty: Impact on Residual Hematoma in a Prospective Controlled Study
Brief Title: Drain Removal Before Versus After CPM in Primary Total Knee Arthroplasty
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Kemal Şibar, Orthopedic Surgeon, Principal Investigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DrainCPM_TKA_2025
Record Dates: First submitted 2025-12-10; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis (Knee OA); Total Knee Anthroplasty; Postoperative Hematoma
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Two-arm prospective parallel-group comparison of drain removal timing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drain Removal Before CPM (Other): The hemovac drain is removed approximately 24 hours after surgery, immediately before a standardized 1-hour CPM session performed at 0-90° flexion. All other perioperative and rehabilitation protocols are identical between groups.
  Interventions: Procedure: Drain Removal Before CPM
- Drain Removal After CPM (Other): Patients undergo a standardized 1-hour CPM session at 0-90° flexion approximately 24 hours after surgery. The hemovac drain is removed immediately after completion of the CPM session. All other perioperative and rehabilitation protocols are identical between groups.
  Interventions: Procedure: Drain Removal After CPM

INTERVENTIONS:
Procedure: Drain Removal Before CPM — Hemovac drain removal performed approximately 24 hours after primary TKA, immediately before a standardized 1-hour CPM session (0-90°). All other surgical, perioperative, and rehabilitation protocols are identical across study arms.
  Arms: Drain Removal Before CPM
Procedure: Drain Removal After CPM — A standardized 1-hour CPM session at 0-90° is administered approximately 24 hours after primary TKA. The hemovac drain is removed immediately after completion of the CPM session. All other surgical, perioperative, and rehabilitation protocols are identical across study arms.
  Arms: Drain Removal After CPM

SUMMARY:
The aim of this prospective randomized controlled study was to determine whether the timing of drain removal in relation to continuous passive motion (CPM) application influences postoperative residual hematoma formation following primary total knee arthroplasty (TKA). Our primary hypothesis was that removing the drain after initiating CPM would result in less residual hematoma, as CPM-induced intra-articular fluid and blood mobilization would be evacuated through the drain before its removal, thereby reducing postoperative fluid accumulation.

DETAILED DESCRIPTION:
This prospective, parallel-group interventional study was conducted at a single tertiary care center between June 2025 and December 2025 following approval by the institutional ethics committee. All patients provided written informed consent prior to participation.

A total of 104 consecutive patients undergoing primary unilateral total knee arthroplasty (TKA) were enrolled during the study period. During follow-up, four patients from each group were lost, leaving 96 patients available for final analysis.

Participants were allocated into two groups using a sequential alternating allocation method (2-1-2-1 sequence). Although not computer-generated, this prospective allocation approach ensured balanced group sizes throughout enrollment. Due to the nature of the intervention, allocation concealment and blinding were not applied.

All surgical procedures were performed by senior arthroplasty surgeons using a standardized medial parapatellar approach under spinal anesthesia. A uniform perioperative protocol was applied to all patients, including antibiotic prophylaxis with intravenous cefazolin and thromboembolism prophylaxis with low-molecular-weight heparin. All procedures were performed under tourniquet control. A single standard intra-articular hemovac drain of identical size and model was placed in all patients prior to wound closure.

Postoperatively, all patients underwent a standardized continuous passive motion (CPM) protocol approximately 24 hours after surgery. CPM was applied for 1 hour with a motion range of 0-90 degrees under supervision of the physiotherapy team.

The only interventional difference between study groups was the timing of drain removal in relation to CPM therapy. In the first group, the hemovac drain was removed immediately before initiation of CPM. In the second group, the drain was removed immediately after completion of the CPM session. All other perioperative care and rehabilitation protocols were identical between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Undergoing primary unilateral total knee arthroplasty (TKA) for end-stage knee osteoarthritis
* Able to provide written informed consent
* Able to comply with scheduled postoperative follow-up assessments

Exclusion Criteria:

* Revision total knee arthroplasty
* Previous infection in the index knee
* Inflammatory arthropathy
* Neuromuscular disorders affecting lower extremity function
* Inability to attend follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2025-06-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Residual Hematoma Formation | Preoperative; Postoperative Day 2; Day 14; Day 28
  Residual hematoma formation assessed by knee circumference measurements at the level of the superior pole of the patella. Circumference is measured on both the operated and contralateral knees. The difference from baseline and between-group differences are evaluated.

SECONDARY OUTCOMES:
Wound Healing | Postoperative Day 2; Day 14
  Wound healing assessed using the Surgical Wound Aspect Score (SWAS), a clinical scoring system evaluating wound characteristics such as swelling (minimum = 0 points, maximum = 2 points), erythema (minimum = 0 points, maximum = 2 points), ecchymosis (minimum = 0 points, maximum = 2 points), blood drainage (minimum = 0 points, maximum = 2 points), and blisters (minimum = 0 points, maximum = 2 points). Finally, a score of 0 points (the best) to 10 points (the worst) was obtained by adding the results of these 5 parameters.
Range of Motion (ROM) | Preoperative; Postoperative Day 2; Day 14; Day 28
  Goniometric measurement of knee flexion and extension on the operated limb. Differences from baseline and between groups are evaluated across postoperative follow-up visits.
Pain Assessment | Preoperative; Postoperative Day 14; Day 28
  Pain intensity assessed using the Visual Analog Scale (VAS), ranging from 0 to 10, where 0 represents no pain and 10 represents the worst imaginable pain. Higher scores indicate greater pain severity.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Preoperative; Postoperative Day 28
  Functional outcome assessed using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), ranging from 0 to 96, where higher scores indicate worse pain, stiffness, and functional limitation.
Lysholm Knee Score | Preoperative; Postoperative Day 28
  Knee function assessed using the Lysholm Knee Score, ranging from 0 to 100, where higher scores indicate better knee function.
Oxford Knee Score | Preoperative; Postoperative Day 28
  Patient-reported knee function assessed using the Oxford Knee Score, ranging from 0 to 48, where higher scores indicate better knee function.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No